CLINICAL TRIAL: NCT03421496
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy, Safety, and Tolerability of Cannabidiol Oral Solution as Adjunctive Therapy With Vigabatrin as Initial Therapy in Patients With Infantile Spasms
Brief Title: A Study to Assess Cannabidiol Oral Solution With Vigabatrin as Initial Therapy in Participants With Infantile Spasms
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to slow enrollment and failure to identify adequate patients that met entry criteria.
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS011-16-082
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Infantile Spasm
Keywords: Infantile spasm; Vigabatrin; Cannabidiol oral solution
MeSH Terms: conditions — Spasms, Infantile | interventions — Cannabidiol; Vigabatrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD with Vigabatrin (Experimental): Participants received up to 40 milligrams per kilogram per day (mg/kg/day) divided twice daily (BID) of CBD with food. Participants also received up to 150 mg/kg/day BID of vigabatrin with food.
  Interventions: Drug: Cannabidiol Oral Solution; Drug: Vigabatrin
- Placebo with Vigabatrin (Placebo Comparator): Participants received a matching placebo to CBD with food, and also received up to 150 mg/kg/day BID of vigabatrin with food.
  Interventions: Drug: Placebo; Drug: Vigabatrin

INTERVENTIONS:
Drug: Cannabidiol Oral Solution — An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).
  Arms: CBD with Vigabatrin
Drug: Placebo — Matching oral solution
  Arms: Placebo with Vigabatrin
Drug: Vigabatrin — Powder suspension
  Other Names: Sabril

SUMMARY:
The primary purpose of this study was to evaluate the efficacy, safety, and tolerability of Cannabidiol Oral Solution (CBD) as adjunctive therapy with vigabatrin as initial therapy, compared to vigabatrin alone in the treatment of infants newly diagnosed with Infantile Spasms (IS).

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, parallel-group study in which participants were randomized in a 1:1 ratio to 1 of 2 treatment groups. During the Initial Treatment Period, participants received either vigabatrin plus CBD or vigabatrin plus matching placebo and were dosed approximately every 12 hours, with a meal. This study was comprised of five periods: Screening, Initial Treatment, Extended Treatment, Taper, and Follow up Periods, with a maximum duration of approximately 140 days.

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s)/caregiver(s) fully comprehends and signs the informed consent form, understands all study procedures, and can communicate satisfactorily with the Investigator and study coordinator, in accordance with applicable laws, regulations, and local requirements.
2. Clinical diagnosis of Infantile Spasms, confirmed by video-EEG (including at least one cluster of electroclinical spasms [≥3 in any 10-minute epoch] and hypsarrythmia) obtained during the Screening Period and read by a central reader.
3. General good health (defined as the absence of any clinically relevant abnormalities as determined by the Investigator) based on physical and neurological examinations, medical history, and clinical laboratory values completed during the Screening Visit).
4. In the opinion of the investigator, the parent(s)/caregiver(s) is (are) willing and able to comply with the study procedures and visit schedules.

Exclusion Criteria:

1. Is considered by the investigator, for any reason (including, but not limited to, the risks described as precautions, warnings, and contraindications in the current version of the Investigator's Brochure for Cannabidiol Oral Solution) to be an unsuitable candidate to receive the study drug.
2. Known or suspected allergy to cannabidiol.
3. History of an allergic reaction or a known or suspected sensitivity to any substance that is contained in the investigational product formulation.
4. Use of any cannabidiol/cannabis product within 30 days of study entry.
5. Participant is diagnosed or suspected of having tuberous sclerosis.
6. Participant has received treatment with either vigabatrin, ACTH, or high-dose steroids previously.
7. Previous or concomitant therapy with felbamate, clobazam, valproic acid, or the ketogenic diet.
8. Participant currently on any disallowed CYP3A4-related medication (phenytoin, fluvoxamine, carbamazepine, and St. John's Wort).
9. Previously received any investigational drug or device or investigational therapy within 30 days before Screening.
10. Clinically significant abnormal laboratory values, including: liver function tests (LFTs) such as albumin, direct bilirubin, total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≥3 times the upper limit of normal (ULN). The investigator may deem the participant eligible if he or she judges the laboratory values to be not clinically significant.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Nicklaus Children's Hospital, Miami, Florida
  - Beaumont Children's Hospital, Royal Oak, Michigan
  - Akron Children's Hospital, Akron, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Institute for Research and Innovation | MultiCare Health System, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Pre-assignment Details: This study was comprised of five periods. The Screening Period lasted up to 14 days, the Initial Treatment period lasted up to 15 days, the Extended Treatment period lasted up to 75 days, followed by a 6-day Taper period and a 30 day Follow up period, with a maximum duration of approximately 140 days.
Groups:
- CBD With Vigabatrin: Participants received up to 40 mg/kg/day twice daily (BID) of CBD orally with food during the 15-day Initial Treatment Period. Participants also received up to 150 mg/kg/day BID of vigabatrin orally with food. During the Extended Treatment Period, complete responders continued their assigned treatment of vigabatrin plus CBD 40 mg/kg/day up to Day 75.
- Placebo With Vigabatrin: Participants received a matching placebo to CBD, orally with food during the 15-day Initial Treatment Period. Participants also received up to 150 mg/kg/day BID of vigabatrin orally with food. During the Extended Treatment Period, complete responders continued their assigned treatment of vigabatrin plus matching placebo up to Day 75.
Period: Overall Study
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Groups:
- CBD With Vigabatrin: Participants received up to 40 mg/kg/day BID of CBD orally with food during the 15-day Initial Treatment Period. Participants also received up to 150 mg/kg/day BID of vigabatrin orally with food. During the Extended Treatment Period, complete responders continued their assigned treatment of vigabatrin plus CBD 40 mg/kg/day up to Day 75.
- Total: Total of all reporting groups
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Considered Complete Responders
Description: Complete response is defined as complete resolution of spasms and hypsarrhythmia confirmed by 24-hour video-electroencephalogram (EEG).
Time Frame: Up to Day 15
Population: as for baseline characteristics
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Resolution of Infantile Spasms
Description: Resolution of IS was assessed by 24-hour video-EEG.
Time Frame: Up to Day 15
Population: as for baseline characteristics
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Resolution of Hypsarrhythmia
Description: Resolution of hypsarrhythmia was assessed by 24-hour video-EEG.
Time Frame: Up to Day 15
Population: as for baseline characteristics
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Investigator Impression of Efficacy and Tolerability of Study Drug Clinical Global Impression- Global Improvement (CGI-I)
Description: Investigators will use the CGI-I scale, which is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and is rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Higher scores indicated worse condition.
Time Frame: Day 15
Population: as for baseline characteristics
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Increase in Number of Spasm-Free Days Between Day 1 and Day 15
Description: Increase in spasm-free days will be determined by seizure diary entries.
Time Frame: Up to Day 15
Population: as for baseline characteristics
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Complete Response During the Initial Treatment Period Who Relapse During the Extended Treatment Period
Description: Relapse during the extended treatment period will be confirmed by video-EEG following parent report of relapse.
Time Frame: Up to Day 75
Population: as for baseline characteristics
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Relapse During the Extended Treatment Period
Time Frame: Up to Day 75
Population: as for baseline characteristics
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Description: This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Arm/Group | CBD With Vigabatrin | Placebo With Vigabatrin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated by the Sponsor. The Sponsor terminated the study due to slow enrollment and a failure to identify adequate participants that met eligibility criteria. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03421496/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03421496/SAP_001.pdf